CLINICAL TRIAL: NCT07185659
Title: The Effect of Walking Exercise on Anxiety, Depression, Dyspnea, Life and Sleep Quality in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: The Effect of Walking Exercise in Patients With Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Pei-Ching Hung, HEAD NURSE, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-XD-098
Record Dates: First submitted 2023-02-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to either the experimental group (E group) or the control group (C group).
  The experimental group received standard care, walking exercise, and elastic band exercise, and wore a smart bracelet to record walking steps and sleep for three months. During the first month, participants performed walking exercise for 100 minutes per week and used a red elastic band for resistance training. In the second month, walking exercise increased to 150 minutes per week with a green elastic band. In the third month, walking exercise increased to 150-300 minutes per week with a blue elastic band.
  The control group wore a smart bracelet to record walking steps and sleep for three months but did not participate in the structured exercise program
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walking exercise and resistance exercise with elastic band (Experimental): From weeks 1 to 12, participants' daily walking steps were monitored using a wearable device (smart bracelet).
  Participants performed walking exercises 5 days per week, twice daily (morning and evening sessions). In weeks 1-4, the prescribed dose was 100 minutes per week (10 minutes per session); in weeks 5-8, 150 minutes per week (15 minutes per session); and in weeks 9-12, 150 to 300 minutes per week (20 to 30 minutes per session).
  Leg resistance extension exercises were also performed with progressively stronger elastic bands: red (weeks 1-4), green (weeks 5-8), and blue (weeks 9-12). During weeks 1-2 and 5-6, exercises were performed 3 times per week with 2 sets per session, which increased to 3 sets per session during weeks 3-4, 7-8, and 11-12.
  Interventions: Device: Elastic band; Device: Xiaomi Mi Band 4 wearable device; Behavioral: Walking
- routine nursing care and health education (Placebo Comparator): Participants received routine nursing care and health education. From weeks 1 to 12, their daily walking steps were monitored using a wearable device (smart bracelet)
  Interventions: Device: Xiaomi Mi Band 4 wearable device

INTERVENTIONS:
Device: Elastic band — Thera-Band® elastic band exercise protocol:
  First stage (weeks 1-4): Participants performed leg resistance stretching exercises with a red elastic band. In weeks 1-2, exercises were performed 3 times per week, with 2 sets per session; in weeks 3-4, 3 times per week, with 3 sets per session.
  Second stage (weeks 5-8): Participants performed leg resistance stretching exercises with a green elastic band. In weeks 5-6, exercises were performed 3 times per week, with 2 sets per session; in weeks 7-8, 3 times per week, with 3 sets per session.
  Third stage (weeks 9-12): Participants performed leg resistance stretching exercises with a blue elastic band. In weeks 9-10, exercises were performed 3 times per week, with 2 sets per session; in weeks 11-12, 3 times per week, with 3 sets per session.
  Arms: walking exercise and resistance exercise with elastic band
Device: Xiaomi Mi Band 4 wearable device — The Xiaomi Mi Band 4 wearable device has been certified by the National Communications Commission (Certification No. CCAG19LP0080T6). From weeks 1 to 12, participants' daily walking steps were monitored using the Xiaomi Mi Band 4 wearable device.
Behavioral: Walking — Walking exercise plan
  Arms: walking exercise and resistance exercise with elastic band

SUMMARY:
"Patients were divided into two groups: the experimental group (E group) and the control group (C group). The E group received standard care, walking exercise, and elastic band exercise, and wore a smart bracelet to record walking steps and sleep for three months. During the first month, participants performed walking exercise for 100 minutes per week and used a red elastic band for resistance training. In the second month, walking exercise increased to 150 minutes per week with a green elastic band. In the third month, walking exercise increased to 150-300 minutes per week with a blue elastic band. The C group wore the smart bracelet to record walking steps and sleep for three months. Each group included 34 participants. The study was conducted from September 9, 2021, to December 31, 2025. Exclusion criteria included panic disorder, cognitive impairment, current cancer treatment, angina pectoris or myocardial infarction within the past 3 months, participation in high-intensity rehabilitation exercise, and walking dysfunction. Participants were required to follow the study protocol.

* Assessments**:
* Anxiety and Depression**:Measured using the Chinese version of the Hospital Anxiety and Depression Scale (HADS).
* Dyspnea**:Measured using the Modified Medical Research Council (mMRC) scale.
* Life and Sleep quality**:Measured using the COPD Assessment Test (CAT) and Chinese Version of the Pittsburgh Sleep Quality Index (CPSQI).

DETAILED DESCRIPTION:
Patients will be divided into two groups: the experimental group (E group) and the control group (C group).

The E group will receive standard care, walking exercise, and elastic band exercise, and will wear a smart bracelet to record walking steps and sleep for three months. During the first month, participants will perform walking exercise for 100 minutes per week and use a red elastic band for resistance training. In the second month, walking exercise will increase to 150 minutes per week with a green elastic band. In the third month, walking exercise will increase to 150-300 minutes per week with a blue elastic band.

The C group will wear a smart bracelet to record walking steps and sleep for three months.

Each group will enroll 34 participants. The study period is from September 9, 2021, to December 31, 2025. Participants with contraindications such as panic disorder, cognitive impairment, ongoing cancer treatment, angina pectoris or myocardial infarction within the past 3 months, participation in high-intensity rehabilitation exercise, or walking dysfunction will be excluded at enrollment based on the exclusion criteria. Participants are required to follow the study protocol.

ELIGIBILITY:
Participants were recruited according to the following criteria.

Inclusion Criteria:

* Inpatients diagnosed with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
* Age ≥ 40 years.
* Post-bronchodilator FEV₁/FVC ratio < 70%.
* History of smoking.
* Ability to perform walking exercises.
* Willingness of the patient or a family member to provide written informed consent.

Exclusion Criteria:

* Panic disorder.
* Presence of delirium with inability to cooperate.
* Currently receiving cancer treatment.
* Angina pectoris or myocardial infarction within the past 3 months.
* Currently undergoing high-intensity rehabilitation exercises.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Patients were assessed before discharge as the baseline, and reassessed at 4, 8, and 12 weeks post-discharge.
  HADS was used to assess differences between groups and over time. The questionnaire consists of 14 items: 7 for anxiety and 7 for depression. Scores range from 0 to 21 for each subscale, with higher scores indicating greater levels of anxiety and depression.
modified Medical Research Council (mMRC) | Patients were assessed before discharge as the baseline, and reassessed at 4, 8, and 12 weeks post-discharge.
  The mMRC scale was used to assess differences in dyspnea severity between groups over time. The mMRC is a five-point scale ranging from 0 (least severe) to 4 (most severe), with higher scores indicating greater dyspnea severity.
COPD Assessment Test (CAT) | Patients were assessed before discharge as the baseline, and reassessed at 4, 8, and 12 weeks post-discharge.
  The COPD Assessment Test (CAT) was used to assess differences between groups over time. The CAT consists of 8 items scored from 0 to 5, yielding a total score of 0 to 40, with higher scores indicating a greater impact of COPD on quality of life.
Chinese Version of the Pittsburgh Sleep Quality Index (CPSQI) | Patients were assessed before discharge as the baseline, and reassessed at 4, 8, and 12 weeks post-discharge.
  CPSQI was used to assess differences between groups over time. Scores range from 0 to 21, with higher scores indicating poorer sleep quality. A score greater than 5 denotes poor sleep quality.
Six-Minute Walk Test ( 6MWT ) | Patients were assessed before discharge as the baseline, and reassessed at 4, 8, and 12 weeks post-discharge.
  The six-minute walk test (6MWT) was used to assess differences between groups and over time. It is an important measure of patients' functional exercise capacity.

SECONDARY OUTCOMES:
Daily walking activity:(1)total steps | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  The Xiaomi Mi Band 4 wearable device will be used to measure daily walking activity, including total steps. Data will be collected to compare differences between two groups over time. By analyzing changes in walking activity over a 12-week period, the effectiveness of the therapeutic intervention will be evaluated.
Daily walking activity:(2)total walking distance | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  The Xiaomi Mi Band 4 wearable device will be used to measure daily walking activity, including total walking distance. Data will be collected to compare differences between two groups over time. By analyzing changes in walking activity over a 12-week period, the effectiveness of the therapeutic intervention will be evaluated.
Sleep status : (1)daily total sleep duration | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  Daily total sleep duration (in hours) was measured using the Xiaomi Mi Band 4 wearable device. The data were collected to evaluate between-group differences and temporal changes. The effectiveness of the therapeutic intervention was investigated by comparing differences in sleep status over 12 weeks.
Sleep status : (2)daily light sleep duration | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  Daily light sleep duration (hours) was measured using the Xiaomi Mi Band 4 wearable device. Data were collected to assess between-group differences and temporal changes. The effectiveness of the therapeutic intervention was evaluated by examining changes in sleep status over 12 weeks.
Sleep status : (3) Daily deep sleep duration | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  Daily deep sleep duration (hours) was measured using the Xiaomi Mi Band 4 wearable device. Data were collected to assess between-group differences and temporal changes. The effectiveness of the therapeutic intervention was evaluated by examining changes in sleep status over 12 weeks.
Sleep status : (4) the number of awakenings during sleep | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  The number of awakenings during sleep was measured using the Xiaomi Mi Band 4 wearable device. Data were collected to assess between-group differences and temporal changes. The effectiveness of the therapeutic intervention was evaluated by examining changes in sleep status over 12 weeks.
Sleep status : (5) total wake time during sleep | Patients were monitored over a 12-week period, with formal assessments conducted at 4, 8, and 12 weeks post-discharge.
  Total wake time during sleep was measured using the Xiaomi Mi Band 4 wearable device. Data were collected to assess between-group differences and temporal changes. The effectiveness of the therapeutic intervention was evaluated by analyzing longitudinal changes in sleep status over 12 weeks."

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ching Hung, Hand nurse, Principal Investigator — Taipei Tzuchi hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Xindian Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No
Protecting participant privacy is the primary consideration, as sharing individual participant data (IPD) could expose sensitive information and create risks of re-identification, even after de-identification. Moreover, participants did not provide consent for data sharing, and obtaining re-consent would be difficult. Ensuring data security also requires substantial resources and technical safeguards that exceed our current infrastructure. In addition, compliance with complex legal and ethical regulations governing data sharing further complicates implementation. Finally, maintaining the quality and integrity of IPD prior to sharing demands additional effort and resources. Collectively, these factors inform our decision to prioritize participant protection and data security.